CLINICAL TRIAL: NCT02296619
Title: The Effects of TAP Block on Hemodynamic Variables, Anaesthetic and Analgesic Requirement and Quality of Recovery in Patients Undergoing Total Abdominal Hysterectomy
Brief Title: The Effects of Transversus Abdominis Plane Block in Patients Undergoing Total Abdominal Hysterectomy
Acronym: TAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, assistant professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GaziosmanpashaU
Record Dates: First submitted 2014-11-13; First posted 2014-11-20 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Abdominal Hysterectomy (& Wertheim); Intraoperative Complications
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP Block (Experimental): Using real time ultrasound imaging, bilateral, 20 ml 0,25% bupivacaine inject into the area between the internal oblique and transverse abdominis muscle
  Interventions: Procedure: TAP block
- Control (Sham Comparator): A sham band-aid will be applied to the abdomen of subjects who are randomized to the no intervention group.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: TAP block — Using real time ultrasound imaging, bilateral, 20 ml 0,25% bupivacaine inject into the area between the internal oblique and transverse abdominis muscle
  Other Names: Transversus abdominis plane block
  Arms: TAP Block
Procedure: Control — A sham band-aid will be applied to the abdomen of subjects
  Other Names: sham group
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effects of Transversus Abdominis Plane Block on hemodynamic variables, anaesthetic and analgesic requirement, and quality of recovery in patients undergoing total abdominal hysterectomy

DETAILED DESCRIPTION:
Pain is one of the main causes of the poor perioperative outcomes and pain management is the important part of perioperative period. Neuraxial blocks could provide adequate analgesia during and after abdominal surgery. However,neuraxial blocks have a lot of contraindicated situations and neuraxial anesthesia can easily induce hemodynamic abnormalities. Therefore, in most cases, the choice of anaesthetic management may be the general anesthesia. In addition to reduce the blood pressure and heart rate changes due to surgical stimulations, the large amount of opioids and anaesthetics may be required. Opioid related side effects can affect perioperative complications and postoperative quality of recovery. Transversus abdominis plane block is a new choice to reduce postoperative pain in abdominal surgery. Although its postoperative analgesic efficacy is well known, its effects on hemodynamic variables, anaesthetic and analgesic requirement is not clear. The main objective of this study is to estimate the effect of Transversus abdominis plane block on hemodynamic variables, anaesthetic and analgesic requirement and quality of recovery in patients undergoing total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-65years old)
* American Society of Anesthesiologists (ASA) physical status I-II
* Patients scheduled for elective total abdominal hysterectomy under general anesthesia

Exclusion Criteria:

* ASA physical status ≥ 3
* Allergy to local anesthetics
* Drug abuse or addiction
* Bleeding tendency

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
intraoperative opioid consumption | during anaesthesia
  The overall intravenous remifentanyl consumption (microgram/ kilogram) during the surgery. The decision to administer remifentanyl is guided by the changes of blood pressure and/ or heart rate greater than 20% from baseline level.

SECONDARY OUTCOMES:
Quality of recovery | postoperative 24 hours
  quality of recovery 40 form will use to assessment the recovery
Postoperative nausea and vomiting | postoperative 0.,2.,12.,24 hours
  nausea score(0-3) and number of vomiting will be recorded
postoperative pain | postoperative 0,2,12,24 hours
  visual analog scale will be used
intraoperative hemodynamic variables | during anaesthesia
  arterial blood pressure, heart rate changes will be recorded
intraoperative anaesthetic consumption | during anaesthesia
  anaesthetic consumption will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Karaman, MD, Principal Investigator — GOU
Locations (1):
- Gaziosmanpasa University Hospital, Tokat Province, Merkez, Turkey (Türkiye)